CLINICAL TRIAL: NCT05070325
Title: Shotblocker or Cold Application; Which One is More Effective in Reducing the Pain Associated With the Intramuscular Injection in Children: A Randomized Controlled Trial
Brief Title: Nonpharmacological Methods for Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bandırma Onyedi Eylül University (Other)
Responsible Party: Principal Investigator, Diler Yilmaz, PhD, RN, Associate Professor, Bandırma Onyedi Eylül University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: BANU-D-YILMAZ-001
Record Dates: First submitted 2021-09-16; First posted 2021-10-07 (Actual); Last update posted 2021-10-15 (Actual); Status verified 2021-10

CONDITIONS: Child; Procedural Anxiety; Procedural Pain
Keywords: Cold application; Intramuscular injection; Pediatric nurse; Shotblocker
MeSH Terms: conditions — Pain, Procedural | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Prospective, randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cold application group (Group 1) (Experimental): In the children in this group, the injection site was cleaned before the injection using antiseptic cotton and then the gel pad was placed on the injection site. In line with the literature, the cold gel pad was applied to the intramuscular injection site for 30-45 seconds before the injection and then the injection was delivered. The children were told to breathe deeply and not to tense up during the injection.
  Interventions: Other: Cold application group
- Shotblocker group (Group 2) (Experimental): The injection site was cleaned using antiseptic cotton. The surface of the Shotblocker with the contact points was placed on the site just before the injection in a way not to contaminate the injection point. Injection was carried out through the opening in the middle of ShotBlocker. The children were told to breathe deeply and not to tense up during the injection. After the injection was completed, ShotBlocker was removed from the skin.
  Interventions: Other: Shotblocker group
- Control Group (Group 3) (Experimental): The routine IM injection was applied to the children in this group. The injection site was cleaned using antiseptic cotton. The children were told to breathe deeply and not to tense up during the injection.
  Interventions: Other: Control Group

INTERVENTIONS:
Other: Cold application group — Cold application group (Group 1): In the children in this group, the injection site was cleaned before the injection using antiseptic cotton and then the gel pad was placed on the injection site. In line with the literature, the cold gel pad was applied to the intramuscular injection site for 30-45 seconds before the injection and then the injection was delivered. The children were told to breathe deeply and not to tense up during the injection.
  Arms: Cold application group (Group 1)
Other: Shotblocker group — Shotblocker group (Group 2): The injection site was cleaned using antiseptic cotton. The surface of the Shotblocker with the contact points was placed on the site just before the injection in a way not to contaminate the injection point. Injection was carried out through the opening in the middle of ShotBlocker. The children were told to breathe deeply and not to tense up during the injection. After the injection was completed, ShotBlocker was removed from the skin.
  Arms: Shotblocker group (Group 2)
Other: Control Group — Control Group (Group 3): The routine IM injection was applied to the children in this group. The injection site was cleaned using antiseptic cotton. The children were told to breathe deeply and not to tense up during the injection.
  Arms: Control Group (Group 3)

SUMMARY:
The study was designed as a randomized controlled experimental research with the purpose of determining the effect of the methods of cold application and Shotblocker on the pain and anxiety level of the children in reducing the pain associated with the intramuscular injection.

The hypotheses of the study:

Hypothesis 0. Shotblocker and the cold application to the injection site prior to the injection are not effective in reducing the pain associated with the intramuscular injection in children.

Hypothesis 1. Using ShotBlocker during the intramuscular injection reduces the pain and anxiety experienced by the child.

Hypothesis 2. Applying cold to the injection site prior to the intramuscular injection reduces the pain and anxiety experienced by the child.

This research was designed as a randomized controlled experimental study in a university hospital in Çorum.

The sample of the study comprised 150 children aged 7 to 12 years who were brought to the pediatric injection room in a university hospital and had intramuscular injection. The children were randomized into the Shotblocker (n=50), cold application (n=50) and control (n=50) groups. In addition to Wong-Baker Pain Scale and Child Anxiety Scale, the Child Information Form was used in the study to determine the introductory characteristics of the children and their family.

DETAILED DESCRIPTION:
The population of this study consisted of the children within the age range of 7-12 years who applied to the injection room in the pediatrics clinic of a university hospital between November 2017 and June 2018. On the other hand, the sample of this study consisted of 150 children who met the case-selection criteria and agreed to participate in the study.

In the Power analysis carried out based on the literature, the sample size of the study was determined as 150 with the confidence level of 90% (α=0.10). For 150 children, the power was β=0.20, 1-β=0.80 with α =.05. The approximate number of subjects was calculated as 50 per group with the Cohen's effect size of α = .05 and the confidence interval of 95%. The children in the sample were randomly assigned to the following groups: Cold application, Shotblocker, and control. In order to determine which case to include in which group, the numbers were randomly distributed to the 3 groups without repetition using a software. In the study, the sample size for each of the 3 groups, that is, cold application group (n=50), Shotblocker group (n=50), and control group (n=50) was determined as 50.

The intramuscular injection was carried out in the pediatric injection room of a university hospital. Before the intervention, the parents and children were met, they were informed about the study, and they were asked whether they would accept to participate in the study. The written and verbal consent were obtained from the parents and the children, respectively. In order to ensure reliability in the study results, the intramuscular injection was applied by the same nurse having at least 5 years of working experience throughout the study; and the pain behavior and anxiety levels of the children were evaluated by the same researcher. The parents were allowed to stay with their children during the intramuscular injection.

The following information was obtained from the children and parents who agreed to participate in the study using the Child Information Form: the socio-demographic characteristics of the children and parent, the previous history of IM injection, the previous history of being subject to a painful intervention, whether the child took an analgesic drug within the last 6 hours, the body mass index (BMI), etc. Prior to the intramuscular injection, the children's weight and height were measured and recorded. The same medicine (procaine penicilline) was administered to all children.

During the intramuscular injection, it was ensured that the environmental factors (temperature, light, noise, etc.), the injection site, and the antiseptic solution (70% alcohol) were standardized. The injection site was wiped using an antiseptic (batticon/chlorhexidine) cotton by gently pressing from center to periphery. It was ensured that the child was in the appropriate position, that is, in the prone position, with the toes facing inward. Prior to the injection, Shotblocker or the cold gel pad was introduced to the children in the experimental group and they were informed of how they would be used. Furthermore, the children and parents were informed about the Wong-Baker FACES® Pain Rating Scale and Children's Fear Scale (CFS) to be used in the study. The parents and children who volunteered to take part in the study were informed of the scale scoring. Which parent would take part in the study was left to the choice of parents to take participate. The CFS scale was evaluated preoperatively after receiving consent from the children and parents and completing the information form. The pain evaluation was made by the children, parents, and observers right after the procedure. When applying the scales, a particular attention was paid so that the children, parents and observers would not see each other's evaluation and not affect one another. Before the injection, the anxiety level was evaluated by the child, parent, and researcher using Children's Fear Scale (CFS). After the injection; the pain level was evaluated by the child, parent, and researcher using the Wong-Baker FACES® Pain Rating Scale, and the anxiety level was evaluated by the parent and researcher using Children's Fear Scale (CFS).

The data of the study was collected using the Child Information Form, the Wong-Baker FACES® Scale, and Children's Fear Scale.

Child Information Form: This form was prepared by the researcher to get information about the children selected for the sample. This form contains a total of 12 questions such as socio-demographic characteristics of the children, whether the child has a health problem that affects her/his perception of pain, the previous history of IM injection, injection duration, and whether the child has injection fear, etc.

Wong-Baker FACES® Scale (WB-FACES): In this scale, there are six faces representing the pain in an increasing order of intensity from zero to five from left to right. The leftmost face has a smile on it, representing "no pain"; whereas the rightmost face has a crying expression, representing "the most intense pain." As the score obtained from the scale increases, the pain tolerance decreases, and vice versa. In practice, the child is asked to choose the face that best expresses her/his feelings. In the application of the scale, it is explained to the child that each face belongs to a person, and the faces represent a happy person with no pain or a sad person feeling a little or too much pain.

Children's Fear Scale (CFS): The scale is used to measure the levels of fear and anxiety in children. The child is shown a picture of 5 facial expressions, each having a score between "0" and "4" points. This scale can be easily applied by both researchers and families to measure the fear and anxiety before and during the applications. In the scale, while "0" refers to "no fear and anxiety"; "4" refers to "the highest fear and anxiety".

The data obtained in this study was analyzed using IBM SPSS Statistics 22 (IBM SPSS, Turkey). The fitness of the parameters to normal distribution was evaluated by the Shapiro-Wilks test. In the evaluation of the data, in addition to the descriptive statistical methods (Mean, Standard deviation, Frequency), one-way analysis of variance (ANOVA) test was used for the comparisons of three or more groups with normal distribution and Tamhane's T2 for the paired comparisons. On the other hand, Chi-Square test was used for the comparison of the qualitative data. The statistical significance was set at p<0.05.

Permission was obtained from the clinical research ethics committee (29.07.16 / 2016-41) to implement the study, and from the relevant institution to carry out the study. Before starting the research, all the children and parents were informed of the purpose of the study, how the study would be carried out, and how the data of the study would be used; and then their verbal and written consent were obtained through the Voluntary Informed Consent Form. Furthermore, they were informed that they could quit the study at any time without giving any reason.

ELIGIBILITY:
Inclusion Criteria: Children

* were in the age group of 7-12 years
* due to IM injection (penicilline (procaine penicilline)

Exclusion Criteria:

* had developmental retardation/disability
* had communication difficulty
* had no chronic disease
* had a history of analgesic drug within the last 6 hours

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 150 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-12-20 (Actual)

PRIMARY OUTCOMES:
Wong-Baker FACES® Scale | Through painful procedure completion, an average of 10 minutes
  The WB-FACES was developed by Wong and Baker in 1981 and revised in 1983. The scale is used to diagnose pain in children aged 3-18 years. It consists of six facial expressions, each one representing an increasing degree of pain scored on a scale 0 to 5 from left to right (0 = very happy/no pain, 5 = the worst pain imaginable). The first face is a happy face representing "no pain" (0) while the last face is a crying face representing "the worst pain imaginable" (5). Higher scores indicate low pain tolerance. Participants are asked to choose the facial expression that best represents their pain
Children's Fear Scale | Through painful procedure completion, an average of 10 minutes
  The CFS was developed to measure fear and anxiety in children. It consists of five facial expressions that represent a range from neutral (0) to extreme fear (4). Both researchers and family members can use the CFS to measure fear and anxiety in children before and during procedures

CONTACTS AND LOCATIONS:
Overall Officials: Selen OZAKAR AKÇA, PhD, RN, Associate Professor, Study Chair — Hitit University; Havva Nur PELTEK KENDİRCİ, PhD, MD, Associate Professor, Study Chair — Hitit University
Locations (1):
- Hitit University- Hitit Medical Faculty Hospital Pediatrics Clinic, Çorum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hunseler C, Roth B, Pothmann R, Reinhold P. [Intramuscular injections in children]. Schmerz. 2005 Apr;19(2):140-3. doi: 10.1007/s00482-004-0318-2. German. PMID 15004746
- [Background] Aydin E, Avsar G. Examining the effect of "Shotblocker" in relieving pain associated with intramuscular injection. Complement Ther Med. 2019 Dec;47:102192. doi: 10.1016/j.ctim.2019.09.001. Epub 2019 Sep 3. PMID 31779992
- [Background] Sanlialp Zeyrek A, Takmak S, Kurban NK, Arslan S. Systematic review and meta-analysis: Physical-procedural interventions used to reduce pain during intramuscular injections in adults. J Adv Nurs. 2019 Dec;75(12):3346-3361. doi: 10.1111/jan.14183. Epub 2019 Sep 13. PMID 31452229
- [Background] Bilge S, Aydin A, Gun C, Aldinc H, Acar YA, Yaylaci S, Cinar O, Balci V. Comparison of the efficacy of ShotBlocker and cold spray in reducing intramuscular injection-related pain in adults. A prospective, randomized, controlled trial. Saudi Med J. 2019 Oct;40(10):996-1002. doi: 10.15537/smj.2019.10.24322. PMID 31588477
- [Background] Canbulat Sahiner N, Turkmen AS. The Effect of Distraction Cards on Reducing Pain and Anxiety During Intramuscular Injection in Children. Worldviews Evid Based Nurs. 2019 Jun;16(3):230-235. doi: 10.1111/wvn.12359. Epub 2019 Apr 17. PMID 30997744
- [Background] Yilmaz G, Alemdar DK. Using Buzzy, Shotblocker, and Bubble Blowing in a Pediatric Emergency Department to Reduce the Pain and Fear Caused by Intramuscular Injection: A Randomized Controlled Trial. J Emerg Nurs. 2019 Sep;45(5):502-511. doi: 10.1016/j.jen.2019.04.003. Epub 2019 Jun 27. PMID 31257044
- [Background] Birnie KA, Noel M, Chambers CT, Uman LS, Parker JA. Psychological interventions for needle-related procedural pain and distress in children and adolescents. Cochrane Database Syst Rev. 2018 Oct 4;10(10):CD005179. doi: 10.1002/14651858.CD005179.pub4. PMID 30284240
- [Background] Gad RF, Dowling DA, Abusaad FE, Bassiouny MR, Abd El Aziz MA. Oral Sucrose Versus Breastfeeding in Managing Infants' Immunization-Related Pain: A Randomized Controlled Trial. MCN Am J Matern Child Nurs. 2019 Mar/Apr;44(2):108-114. doi: 10.1097/NMC.0000000000000512. PMID 30807328
- [Background] Canbulat Sahiner N, Turkmen AS, Acikgoz A, Simsek E, Kirel B. Effectiveness of Two Different Methods for Pain Reduction During Insulin Injection in Children With Type 1 Diabetes: Buzzy and ShotBlocker. Worldviews Evid Based Nurs. 2018 Dec;15(6):464-470. doi: 10.1111/wvn.12325. Epub 2018 Oct 11. PMID 30307692
- [Background] Sivri Bilgen B, Balci S. The Effect on Pain of Buzzy(R) and ShotBlocker(R) during the Administration of Intramuscular Injections to Children: A Randomized Controlled Trial. J Korean Acad Nurs. 2019 Aug;49(4):486-494. doi: 10.4040/jkan.2019.49.4.486. PMID 31477677
- [Background] ENA Clinical Practice Guideline Committee; ENA Board of Directors Liaisons:; Methodologist:; Staff Liaisons:; Administrative Staff:. Clinical Practice Guideline: Needle-Related or Minor Procedural Pain in Pediatric Patients. J Emerg Nurs. 2019 Jul;45(4):437.e1-437.e32. doi: 10.1016/j.jen.2019.05.015. No abstract available. PMID 31280767
- [Background] Cobb JE, Cohen LL. A randomized controlled trial of the ShotBlocker for children's immunization distress. Clin J Pain. 2009 Nov-Dec;25(9):790-6. doi: 10.1097/AJP.0b013e3181af1324. PMID 19851160
- [Background] Caglar S, Buyukyilmaz F, Cosansu G, Caglayan S. Effectiveness of ShotBlocker for Immunization Pain in Full-Term Neonates: A Randomized Controlled Trial. J Perinat Neonatal Nurs. 2017 Apr/Jun;31(2):166-171. doi: 10.1097/JPN.0000000000000256. PMID 28437308